CLINICAL TRIAL: NCT00145782
Title: The Ebeltoft Health Promotion Project - A Randomized Controlled Trial With Multiphasic Preventive Health Screenings and Discussions in General Practice.
Brief Title: The Ebeltoft Health Promotion Project
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1990/1966; 2001-41-0738 Data Protec. A; 9801336 Medical Res. Council; 22-04-0434 Danish Research Ag
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2005-09-05 (Estimated); Status verified 2005-09

CONDITIONS: Primary Prevention
Keywords: multiphasic screening; primary health care; randomized controlled trial; Risk factors

INTERVENTIONS:
Behavioral: Life style

SUMMARY:
The objective of The Ebeltoft Health Promotion Project is investigate the effect of multiphasic preventive health screenings and discussions with general practitioners of a random population of patients in primary care.

Outcome parameters are the cardiovascular risk profile, number of health care contacts, life years gained, direct costs, i.e. health care costs, and total cost, i.e. including productivity costs.

DETAILED DESCRIPTION:
The Ebeltoft project was designed as a randomized controlled trial in the district of Ebeltoft, Aarhus County, Denmark. All nine general practitioners (GPs) from the four primary care units in the district participated. All patients listed in the primary care units between 30 and 49 years of age by January 1, 1991 (N=3,464) were identified in the Danish Civil Registration system, each Danish resident has a ten digit number, through which personal data can be extracted from the health and social registries. A random selection of 2,030 of the 3,464 persons was sampled for invitation to participate in the study. Those who agreed to participate were randomly divided into one control group and two intervention groups (A and B). Randomization of subjects into control and intervention groups was stratified by primary care unit, sex, age, body mass index (BMI), and cohabitation status as stated by the subjects in the invitation questionnaire. Invited subjects received an invitation questionnaire in September 1991. All subjects who agreed to participate also received questionnaires about their health, health beliefs, and social and demographic status at baseline and after one and five years. Subjects in the two intervention groups were offered a broad (multiphasic) health screening at baseline and after one and five years. After five years all subjects received a questionnaire and an invitation to a health screening and consultation. From December 1, 1991 to October 1, 1997 specially trained laboratory technicians carried out health screenings that included evaluations of cardiovascular, pulmonary, liver and kidney function, endocrine dysfunction, BMI, physical endurance, hearing and sight. Evaluation of cardiovascular function included a calculation of cardiovascular risk score (CRS), giving an estimate of the risk of premature cardiovascular disease for each individual. CRS was based on sex, familial inheritance (number of family members with ischemic heart disease before age 55), tobacco consumption, blood pressure, total serum cholesterol, and BMI.1 Within three weeks of the screenings, all participants received a written letter from their GP explaining the tests. Targeted life style counsels were included in the letter if the test results were outside a predefined range. All subjects who had been informed that they had an elevated or high CRS were encouraged to see their GP, regardless of their intervention status. After the health screenings, the subjects in group B were invited to attend a 45-minute patient centred health consultation with their GP. The health consultations were aimed primarily at discussing lifestyle-related health problems and giving the subject an opportunity to define up to three goals relating to lifestyle changes.

We investigate the impact of the intervention on the cardiovascular risk profile, number of health care contacts, the direct and total costs, and the health effects by comparing mean costs and expected life years gained of the intervention groups with those of the control group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30 to 49 1. january 1991
* Registered with a local general practitioner in the district of Ebeltoft

Exclusion Criteria:

* Unable to understand and respond to a mailed invitation questionnaire

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 1991-09; Study Completion 1999-12

PRIMARY OUTCOMES:
Cardiovascular risk profile after 5 and 15 years
Life years gained and cost effectiveness after 6 years
All cause mortality after 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Lauritzen, Professor, Study Chair — Institute of Public Health, Dept. of general Practice, University of Aarhus
Locations (1):
- Institute of Public Health, Dept. of General Practice, University of Aarhus, Aarhus, Denmark

REFERENCES:
- [Result] Engberg M, Christensen B, Karlsmose B, Lous J, Lauritzen T. General health screenings to improve cardiovascular risk profiles: a randomized controlled trial in general practice with 5-year follow-up. J Fam Pract. 2002 Jun;51(6):546-52. PMID 12100779
- [Result] Thomsen JL, Parner ET, Karlsmose B, Thulstrup AM, Lauritzen T, Engberg M. Effect of preventive health screening on long-term primary health care utilization. A randomized controlled trial. Fam Pract. 2005 Jun;22(3):242-8. doi: 10.1093/fampra/cmi007. Epub 2005 Apr 6. PMID 15814585
- [Derived] Bernstorff M, Deichgraeber P, Bruun NH, Dalsgaard EM, Fenger-Gron M, Lauritzen T. A Randomised Trial Examining Cardiovascular Morbidity and All-Cause Mortality 24 years Following General Health Checks: the Ebeltoft Health Promotion Project (EHPP). BMJ Open. 2019 Oct 28;9(10):e030400. doi: 10.1136/bmjopen-2019-030400. PMID 31662372